CLINICAL TRIAL: NCT05649774
Title: Effects of Taping & Exercise Therapy on Lower Back Musculoskeletal Conditions in Pakistani Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Kiran Arshad, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KArshad
Record Dates: First submitted 2022-11-19; First posted 2022-12-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Lower Back Pain; Musculoskeletal Diseases or Conditions
Keywords: Lower back pain; Non specific lower back pain
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Diseases | interventions — Therapeutics; Myofascial Release Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: The study was a parallel group, four arm superiority trial with 1:1 allocation ratio and balanced randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Myofascial Release (MFR) (Active Comparator): The therapist will place its hands on the T12-L1 levels as well as on the sacrum. A cross handed hold will be performed along the fascia. Then for the gluteus Medius and maximus muscle, the therapist will stand facing the participant's leg and closed to the superior border of participant's pelvis. The therapist will place the palm of the hand on the anterior surface, allowing the fingers to rest on the outer fibers of the gluteal muscles stabilizing the pelvis of the participants. Allow the participant to flex its knee while applying adequate amount of stretch on the hip joint in an open pack position. Hold, wait for the release and stretch again. for tensor fascia Latae, The therapist will place several slightly adducted fingers of its one hand on the superior fibers proximal to the insertion on the anterior superior iliac crest and the thumb as well as the other fingers of the other hand on the distal muscle fibers. Hold, wait for the release and stretch again.
  Interventions: Procedure: Therapy
- Kinesio Taping (KT) (Active Comparator): Lumbar star correction technique was applied. 4 tape I strips will be cut. The paper from the center will be torn. The targeted area will be stretched as tolerated at the lumbar region. The therapist will apply 25% to 35% tension to the strip within the therapeutic zone over the target tissue. End the strip with no tension and activate the adhesive. For the second strip change the posture in order to change the stretch on the tissue, apply the second strip with 25% to 35% tension in the center of the tape and end with no tension. Activate the adhesive. Now flex the trunk and rotate on one side. Apply the third tape strip with 25% to 35% tension in the center of the tape. Apply the fourth tape strip with flexion and rotation on the opposite side again with 25% to 35% tension on the strip.
  The tape will be changed 3 times per week.
  Interventions: Procedure: Taping technique
- Myofascial Release with Taping (MFKT) (Experimental): Same Protocol of MFR followed by KT
  Interventions: Procedure: Therapy with taping
- Placebo Treatment (Sham Comparator): The control group received a sham myofascial release for 40 minutes per treatment session, three times a week for three weeks. The sham myofascial release was applied by gently placing the hands over the same areas treated in the MFR group,without sliding, just enough to maintain contact for the desired time.
  Interventions: Procedure: SHAM

INTERVENTIONS:
Procedure: Therapy — Only Myofascial Release will be provided
  Other Names: Myofascial Release
  Arms: Myofascial Release (MFR)
Procedure: Taping technique — Only Kinesiotaping will be provided
  Other Names: Taping
  Arms: Kinesio Taping (KT)
Procedure: Therapy with taping — Myofascial release will be provided followed by Kinesiotaping
  Other Names: Therapy followed by taping
  Arms: Myofascial Release with Taping (MFKT)
Procedure: SHAM — Placebo Treatment will be given
  Arms: Placebo Treatment

SUMMARY:
Lower back pain has been one of the most frequently occurring musculoskeletal disorder among the females. This act as a global burden and is highly prevalent in our society. This pain can result in life long disability, loss of function and mobility among individuals. The female of the society suffers from lower back pain the most because of the under lying causes, prolong standing and stooping as well as because of hormonal changes in their bodies

DETAILED DESCRIPTION:
After studying the prevalence of the lower back pain among the females of Pakistan, the investogator find the need to assess the type of their pain and find out the best way to ease their pains. The motive was to develop a treatment protocol whose effects last longer and is inexpensive for the management of lower back pain.

Moreover, the investigator decided to study that which treatment protocol is better when compared to another and what is the role of sham treatment when given to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Females who were willing to participate.
* Participants with nonspecific lower back pain will only be included and screened through the screening questionnaire.

Exclusion Criteria:

* Post-menopausal women
* Females with any diagnosed co-morbidity.
* Back pain progressive to any neurological deficit
* Sustained or increased back pain with loss of appetite and unexplained weight loss accompanied with fever, nausea and chills
* With any known spinal or lower back pathology
* Tumor of the spine
* Any underlying diseases of spinal cord (i.e, ankylosing spondylosis, spondolisthesis)
* With any steroid therapy for lower back pain in the past three months
* Any inflammatory rheumatic disease
* Sensitive skin or any skin allergy or dermatological condition
* Any rehabilitative services taken for the lower back pain in the past two months
* Rejection to manual conatct

Ages: 28 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females will be included in the study because lower back pain is highly prevalent among them.
Enrollment: 100 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Lower Back Pain | Change from baseline to week 3
  Numeric Pain Rating Scale
Disability of lower back | Change from baseline to week 3
  Oswestry Disability Index

SECONDARY OUTCOMES:
Range of Motion | Change from baseline to week 3
  Flexion, Extension and Lateral Bending (L and R)
Pain Pressure Threshold | Change from baseline to week 3
  Algometer was used to check the pain pressure threshold of Thoraco lumbar fascia, Gluteus Medius, Gluteus Maximus and Tensor Fascia Latae
Tissue Hardness | Change from baseline to week 3
  Algometer was used to check the tissue hardness of Thoraco lumbar fascia, Gluteus Medius, Gluteus Maximus and Tensor Fascia Latae
Quality of Life of patients with Lower back pain | Change from baseline to week 3
  36-Item Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Arshad, M.Phil, Principal Investigator — University of Karachi
Locations (1):
- Al-Tibri Medical college and hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be collected in the form of distribution of questionnaire to the participants.
  Confidentiality of the participants will be maintained. Consent will be taken form participants before collection of data.